CLINICAL TRIAL: NCT00791167
Title: Evaluation of the Dose Proportionality of Two Dose Strengths (1.5 and 3 mg) of Extended-release Paliperidone After a Single Administration to Healthy Men
Brief Title: A Study of the Dose Proportionality of Extended Release Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR011437
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: Mood Disorders, Antipsychotic drugs; Schizophrenia; Paliperidone ER
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purposes of this study are to evaluate the dose proportionality of 1.5- and 3 mg tablets of paliperidone ER, to document the pharmacokinetics of a 1.5 mg dose of paliperidone ER, and to assess the safety and tolerability of the 1.5- and 3 mg tablets in healthy men.

DETAILED DESCRIPTION:
This is a randomized, open label, single center, single dose, 2 treatment, 2 way crossover study. It consists of 3 phases: A screening phase beginning within 21 days before the first study drug administration; an open label treatment phase consisting of 2 treatment periods (Period 1 and Period 2) during which volunteers will receive a single oral 1.5 or 3 mg dose of study drug; and end of study evaluations upon completion of all the study procedures in Period 2. All volunteers will receive each of the following 2 treatments in random order: Treatment A: One tablet of 1.5 mg paliperidone ER to-be-marketed formulation in the fasted state; Treatment B: One tablet of 3 mg paliperidone ER Phase 3 formulation in the fasted state. Successive study drug administrations will be separated by a washout period of at least 9 days and no more than 21 days. A 1.5-mg dose of paliperidone ER was selected to be studied as the availability of a 1.5-mg tablet would make dose-adjustments across the existing range of doses of paliperidone ER easier in patients with reduced renal function or tolerability issues. Safety and tolerability of the 1.5- and 3 mg tablets of paliperidone ER in healthy men will be monitored throughout the study.

A single oral doses of 1.5 mg and 3 mg paliperidone ER

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ( weight [kg]/height [m2]) of 18 to 30 kg/m2, inclusive
* Have a supine (after 5 minutes rest) blood pressure between 100 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, 12-lead ECG, and the laboratory results of serum chemistry, hematology, and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology, or urinalysis testing are not within the laboratory's reference ranges, the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For renal function tests, the values must be within the normal laboratory reference ranges

Exclusion Criteria:

* Known drug allergy to risperidone, paliperidone, or any of its excipients
* Known history of drug-induced dystonia
* Recent history of alcohol or substance abuse
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic, or immunologic disease
* History of any cancer, with the exception of basal cell carcinoma
* At screening, has signs of autonomic dysfunction as indicated by a sustained decrease of > 20 mmHg in systolic blood pressure or a decrease of >10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <50 bpm) as determined by screening 12-lead ECG
* A positive test result (or history of) for any of the serology tests (hepatitis B and C, and human immunodeficiency virus) at screening
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. Volunteers must agree to refrain from use throughout the study
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements) within 14 days before the first dose of study drug. Exception for acetaminophen (paracetamol) or ibuprofen, which is allowed up to 3 days before first dose of study drug

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2006-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate dose-proportionality of 1.5 and 3-mg tablets of paliperidone ER

SECONDARY OUTCOMES:
To document the pharmacokinetics of a 1.5-mg dose of paliperidone ER in healthy men and to assess the safety and tolerability of the 1.5- and 3 mg tablets of paliperidone ER in healthy men

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the dose proportionality of extended release paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=733&filename=CR011437_CSR.pdf